CLINICAL TRIAL: NCT02187042
Title: EVALUATION OF THE IMPACT OF A THERAPY MANAGEMENT PLATFORM ON THE MANAGEMENT OF PATIENTS SUFFERING FROM ADVANCED/METASTATIC RENAL CELL CARCINOMA AND RECEIVING FIRST LINE TREATMENT WITH SUNITINIB, VERSUS STANDARD FOLLOW-UP
Brief Title: Evaluation Of The Impact Of A Call Center In Management Of Metastatic And/Or Advanced Renal Cell Carcinoma Patients Treated With Sunitinib (Sutent) In First Line
Acronym: RENACALL
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181213; RENACALL (Other: Alias Study Number)
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Results first posted 2019-10-24 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Metastatic/Advanced Renal Cell Carcinoma
Keywords: sunitinib; call center; management of patients; nurses; metastatic renal carcinoma
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Renal Cell | interventions — Call Centers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: Metastatic and/or advanced renal cell carcinoma patients treated with sunitinib in first line and followed by standard care plus call center
  Interventions: Other: Best supportive care; Other: call center

INTERVENTIONS:
Other: Best supportive care — BSC may include medications and supportive measures deemed necessary to palliate disease related symptoms and improve quality of life
Other: call center — Nurses from a call center will call the patients at regular time to help patients in the management of their cancer, with some dietetic advices, medical advices etc.

SUMMARY:
100 patients with metastatic and/or advanced renal cell carcinoma treated with sunitinib (Sutent) will be inclued and followed with standard care plus a call center

Principal assumption : the proportion of patients presenting with at least one grade 3 or 4 AE (whether related to sunitinib or not).

DETAILED DESCRIPTION:
RENACALL is a prospective intermediate care study whose main aim is to evaluate the impact of a therapy management platform on the management of patients suffering from advanced/metastatic renal cell carcinoma and receiving first line treatment with Sutent®.

100 mRCC patients treated receiving first line Sutent® treatment shall be included in the study, and shall benefit both from conventional follow-up and from additional therapy management platform-based follow-up. Platform follow-up shall consist in regular phone calls to accompany patients in their real life home management of their treatment with sunitinib (prevention, advice and guidance of patients towards options)..

ELIGIBILITY:
Inclusion Criteria:

Man or woman aged 18 or over;

* Patient suffering from a/mRCC, receiving sunitinib first-line treatment, as per SPC recommendations;
* Resolution (grade ≤ 1 according to CTCAE version 4.03 of June 2010) of all acute toxic effects due to radiotherapy or surgical procedure prior to initiation of sunitinib;
* Patient who can be monitored for 6 months.
* Female patient of child-bearing age using a form of contraception during treatment with Sunitinib and for at least 28 days after termination of treatment with Sunitinib;
* Patient having signed his/her consent form;
* Patient affiliated with a social security scheme.

Non-inclusion criteria

* Patient participating in a clinical trial during sunitinib treatment;
* Patient managed by a home hospitalisation service during sunitinib treatment;
* Patient taking part in therapeutic education programmes, or benefiting from nursing consultation, or from any other significant treatment support and likely to impact adverse event management.
* Patient untreated and/or symptomatic brain metastases prior to sunitinib initiation;
* Patient refusing the use of his/her personal data.
* Patient with an ECOG performance status upon inclusion > 2;
* Patient presenting with a serum creatinine level >1.5 times the upper limit of the normal level;
* Patient presenting with a bilirubin level > 2 mg/dl, aspartate transaminase (ASAT) or alanine transaminase (ALAT) >2.5 times the upper limit of the normal value, or >5 times the upper limit of the normal value in the presence of liver metastases upon initiation of sunitinib treatment.
* Patients who are staff members of a centre involved in the study, or close to one of the staff members of a centre directly involved in conducting the study, or patients employed by Pfizer and involved in conducting the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The 100 metastatic and/or advanced patients of the study will come from the population of patients under the care of French renal cell carcinoma oncologists
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2015-10-07 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- France (13):
  - CHU de la Timone, Marseille, Cedex 5
  - CHU Strasbourg, Strasbourg, Cedex
  - Centre Hospitalier d'Annecy, Annecy
  - Centre Catalan Urologie Andrologie, Cabestany
  - Centre hospitalier de Chambery, Chambéry
  - Hopital prive La Louviere, Lille
  - Clinique Claude Bernard Chimiotherapie Ambulatoire, Metz
  - CRLC Val d'Aurelle, Montpellier
  - Polyclinique Gentilly, Nancy
  - Polyclinique de Gentilly Service Oncologie Médicale, Nancy
  - CHI de Cornouailles - Oncologie hospitalisation, Quimper
  - Hopital Jean BERNARD - Tours - 7eme etage, Valenciennes
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181213&StudyName=Evaluation%20Of%20The%20Impact%20Of%20A%20Call%20Center%20In%20Management%20Of%20Metastatic%20And/Or%20Advanced%20Renal%20Cell%20Carcinoma%20Patients%20Treated%20With%20Sunit

RESULTS

PARTICIPANT FLOW:
Groups:
- Call Center: Participants with advanced/metastatic renal cell carcinoma (a/mRCC) being treated first line with sunitinib (dose as per the recommendations in the summary or product characteristics [SmPC]) were followed up conventionally and by call center. Participants were conventionally monitored at the end of Cycles 1, 2 and 4 of sunitinib treatment as routine consultation visit at the oncology care centers. In addition, the follow-up consisted of regular phone calls by the call center nurses using a computer-assisted telephone interview system; participants received 5 calls on Week 1, 2, 3, 4 and 5 of each Cycle 1 and 2 of sunitinib treatment and 2 calls on Week 2 and 4 of each Cycle 3 and 4 of sunitinib treatment. Each cycle was of at least 6 weeks.
- Standard of Care: Participants with a/mRCC being treated first line with sunitinib (dose as per SmPC) were followed by conventional standard care method. Participants were monitored at the end of Cycles 1, 2 and 4 of sunitinib treatment as routine consultation visit at the oncology care centers. Each cycle was of at least 6 weeks.
Period: Overall Study
Arm/Group | Call Center | Standard of Care
Started | 42 | 27
Completed | 29 | 13
Not Completed | 13 | 14
Not completed — Death | 1 | 1
Not completed — Toxicity | 6 | 5
Not completed — Participant choice | 1 | 0
Not completed — Doctor choice | 1 | 0
Not completed — Progressive disease | 4 | 8

BASELINE CHARACTERISTICS:
Population: Safety population included participants treated with Sunitinib.
Groups:
- Call Center: Participants with a/mRCC being treated first line with sunitinib (dose as per the recommendations in the SmPC) were followed up conventionally and by call center. Participants were conventionally monitored at the end of Cycles 1, 2 and 4 of sunitinib treatment as routine consultation visit at the oncology care centers. In addition, the follow-up consisted of regular phone calls by the call center nurses using a computer-assisted telephone interview system; participants received 5 calls on Week 1, 2, 3, 4 and 5 of each Cycle 1 and 2 of sunitinib treatment and 2 calls on Week 2 and 4 of each Cycle 3 and 4 of sunitinib treatment. Each cycle was of at least 6 weeks.
- Total: Total of all reporting groups
Arm/Group | Call Center | Standard of Care | Total
Number analyzed (Participants) | 42 | 27 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (10.3) | 65.6 (9.2) | 66.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 17
  Male | 30 | 22 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least 1 Adverse Event (AE) of Grade 3 or 4 Based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life threatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. The severity was graded by NCI CTCAE v.4.03. Grade 1 was mild AE. Grade 2 was moderate AE. Grade 3 was severe AE. Grade 4 was life-threatening consequences and urgent intervention AE. Grade 5 was death related to AE.
Time Frame: Baseline up to 6 months
Population: Safety population included participants treated with Sunitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Call Center | Standard of Care
Number analyzed (Participants) | 42 | 27
Participants | 34 | 14

2. Secondary Outcome: Number of Participants With at Least 1 Sunitinib Dose Reduction
Description: Number of participants treated with sunitinib having had at least 1 dose reduction relative to the initial dose are reported.
Time Frame: Baseline up to 6 months
Population: Safety population included participants treated with Sunitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Call Center | Standard of Care
Number analyzed (Participants) | 42 | 27
Participants | 12 | 4

3. Secondary Outcome: Number of Participants Involved in at Least 1 Occasion For Each of the Reasons for a Sunitinib Dose Reduction
Description: Number of participants treated with sunitinib having had at least 1 dose reduction relative to the initial dose according to the reasons for dose reductions are reported.
Time Frame: Baseline up to 6 months
Population: Safety population included participants treated with Sunitinib. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Call Center | Standard of Care
Number analyzed (Participants) | 12 | 4
Participants
  Adverse Event | 12 | 3
  Unknown | 0 | 1

4. Secondary Outcome: Average Sunitinib Dose Reduction
Time Frame: Baseline up to 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milligram per day (mg/day)
Arm/Group | Call Center | Standard of Care
Number analyzed (Participants) | 12 | 4
milligram per day (mg/day) | 12.5 (0) | 12.5 (0)

5. Secondary Outcome: Number of Participants With at Least 1 Temporary Interruption of Sunitinib Treatment
Description: Reason for temporary dose interruptions included: who had AEs that were intolerable, surgery, omission, doctor choice and any other reason judged by doctor.
Time Frame: Baseline up to 6 months
Population: Safety population included participants treated with Sunitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Call Center | Standard of Care
Number analyzed (Participants) | 42 | 27
Participants | 27 | 8

6. Secondary Outcome: Mean Duration (in Days) of Temporary Interruption to Sunitinib Treatment
Description: as for outcome 5
Time Frame: Baseline up to 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Call Center | Standard of Care
Number analyzed (Participants) | 27 | 8
days | 10.5 (11.5) | 16.6 (19.4)

7. Secondary Outcome: Number of Participants Involved on at Least 1 Occasion for Each of the Reasons for a Sunitinib Temporary Treatment Interruption
Description: Reason for temporary dose interruptions included: who had AEs that were intolerable, surgery, omission, doctor choice and any other reason judged by doctor. Participants were counted in more than 1 category.
Time Frame: Baseline up to 6 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Call Center | Standard of Care
Number analyzed (Participants) | 27 | 8
Participants
  AE | 19 | 7
  Surgery | 1 | 0
  Omission | 4 | 0
  Doctor choice | 6 | 1
  Other | 2 | 1

8. Secondary Outcome: Number of Participants Who Permanently Discontinued Sunitinib Treatment
Description: Reason for permanent discontinuation of sunitinib treatment included: progressive disease, toxicity, participant's choice, doctor's choice and death of participant.
Time Frame: Baseline up to 6 months
Population: Safety population included participants treated with Sunitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Call Center | Standard of Care
Number analyzed (Participants) | 42 | 27
Participants | 13 | 14

9. Secondary Outcome: Number of Participants Involved on At Least 1 Occasion for Each of the Reasons for a Permanent Sunitinib Treatment Discontinuation
Description: as for outcome 8
Time Frame: Baseline up to 6 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Call Center | Standard of Care
Number analyzed (Participants) | 13 | 14
Participants
  Progressive Disease | 4 | 8
  Toxicity | 6 | 5
  Participant Choice | 1 | 0
  Doctor's Choice | 1 | 0
  Death | 1 | 1

10. Secondary Outcome: Mean Duration of Sunitinib Treatment
Description: Total mean duration (in months) of sunitinib treatment is reported in this outcome measure.
Time Frame: Baseline up to 6 months
Population: Safety population included participants treated with Sunitinib.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Call Center | Standard of Care
Number analyzed (Participants) | 42 | 27
Months | 4.8 (1.9) | 4.2 (1.9)

11. Secondary Outcome: Number of Participants Classified on the Basis of Number of Sunitinib Treatment Cycles
Description: Last treatment cycle was declared by doctor either on the notified date to discontinue sunitinib or on the date of the last consultation if sunitinib treatment was not stopped
Time Frame: Baseline up to 6 months
Population: Safety population included participants treated with Sunitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Call Center | Standard of Care
Number analyzed (Participants) | 42 | 27
Participants
  1 Cycle | 6 | 3
  2 Cycles | 1 | 7
  3 Cycles | 7 | 5
  4 Cycles | 28 | 12

12. Secondary Outcome: Number of Participants With At Least 1 Unplanned Hospitalization
Description: Number of participants with at least 1 unplanned hospitalizations either related or unrelated to sunitinib were reported.
Time Frame: Baseline up to 6 months
Population: Analysis population included participants who were treated with Sunitinib and had follow up by call center along with conventional method. Data was collected only for the reporting arm "call center" as per the planned analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Call Center
Number analyzed (Participants) | 42
Participants | 9

13. Secondary Outcome: Number of Participants With At Least 1 Unplanned Consultation
Description: Number of participants with at least 1 unplanned consultations either related or unrelated to sunitinib were reported.
Time Frame: Baseline up to 6 months
Population: Analysis population included included participants who were treated with sunitinib and had follow up by call center along with conventional method. Data was collected only for the reporting arm "call center" as per the planned analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Call Center
Number analyzed (Participants) | 42
Participants | 16

14. Secondary Outcome: Number of Participants Who Were "Adherent" as Per 4- Item Morisky Medication Adherence Scale (MMAS-4)
Description: MMAS-4 is a self-reported measure of medication taking behavior, consisting of 4 questions based on forgetting taking medication, carelessness about taking medication, stopping medication when feeling better, or stopping medication when feeling worse. Each question has answer either "Yes" or "No"; "Yes" =1 and "No" =0. The sum of answer to all 4 questions resulted in total MMAS-4 score. Total MMAS-4 score ranges from 0 (best adherence) to 4 (worst adherence), a low score representing improved adherence. Adherent participants were defined as participants with an MMAS-4 score of 0.
Time Frame: Baseline up to 6 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Call Center | Standard of Care
Number analyzed (Participants) | 34 | 18
Participants | 30 | 15

15. Secondary Outcome: Mean 4-Item Morisky Medication Adherence Scale (MMAS-4) Score
Description: MMAS-4 is a self-reported measure of medication taking behavior, consisting of 4 questions based on forgetting taking medication, carelessness about taking medication, stopping medication when feeling better, or stopping medication when feeling worse. Each question has answer either "Yes" or "No"; "Yes" =1 and "No" =0. The sum of answer to all 4 questions resulted in total MMAS-4 score. Total MMAS-4 score ranges from 0 (best adherence) to 4 (worst adherence), a low score representing improved adherence. High adherence: score of 0, average adherence: score of 1 or 2, poor adherence: score of 3 or 4.
Time Frame: Baseline up to 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Call Center | Standard of Care
Number analyzed (Participants) | 34 | 18
Units on a scale | 0.1 (0.5) | 0.2 (0.4)

16. Secondary Outcome: Objective Response Rate (ORR): Percentage of Participants With a Complete or Partial Best Response
Description: ORR used for the assessment of response to treatment. As per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1: Complete response (CR) was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis less than [<] 10 millimetre [mm]). No new lesions. Partial response (PR) was defined as greater than or equal to (>=) 30 percent (%) decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: Baseline up to 6 months
Population: Analysis population included all participants who were investigated by the doctors, who met the study eligibility criteria, had received at least 1 dose of Sunitinib and who had telephone calls with call center. Data was collected only for the reporting arm "call center" as per the planned analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Call Center
Number analyzed (Participants) | 39
Percentage of participants | 33.3

17. Secondary Outcome: Mean Scores for Each Dimension on the Participant's Satisfaction (With the Management By the Telephone Call Center) Questionnaire
Description: Participants' satisfaction with call center was assessed via the self-administered questionnaire completed at the end of the study. Questionnaire evaluated 4 dimensions with total of 8 items. Dimensions were: 1) Satisfaction with advice: 3 item, 2) Satisfaction with care, 3) Satisfaction concerning the service: 3 items and 4) Overall satisfaction with support in management of sunitinib treatment: 1 item. Each item had 5 responses: very satisfied, satisfied, not very satisfied, not satisfied and no opinion equivalent to score of +2, +1, 1, -2 and no score respectively. A score was calculated for each dimension by calculating the mean scores obtained for each item if at least 50% of the items for the dimension had been completed (and are not "no opinion"). Overall possible mean score range for each dimension was +2 to -2, where higher scores signified higher satisfaction.
Time Frame: At the end of the study (At Month 6)
Population: Analysis population: participants who were investigated by the doctors, who met study eligibility criteria, had received at least 1 dose of Sunitinib and were followed up by call center and completed a self-administered satisfaction questionnaire about management by call center. Here, 'Number analyzed' = participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Call Center
Number analyzed (Participants) | 22
Units on a scale
  Satisfaction with the advice: number analyzed (Participants) | 21
  Satisfaction with the advice | 1.2 (0.9)
  Satisfaction with care: number analyzed (Participants) | 21
  Satisfaction with care | 1.1 (1.1)
  Satisfaction with the service: number analyzed (Participants) | 19
  Satisfaction with the service | 1.2 (0.9)
  Overall satisfaction with support in management: number analyzed (Participants) | 21
  Overall satisfaction with support in management | 1.2 (0.9)

18. Secondary Outcome: Number of Participants Who Reported Themselves Being "Satisfied" or "Very Satisfied" With the Management By the Telephone Call Center
Description: Participants' satisfaction with call center was assessed via the self-administered questionnaire completed at the end of the study. Questionnaire evaluated 4 dimensions with total of 8 items. Dimensions were: 1) Satisfaction concerning advice: have 3 item, 2) Satisfaction concerning management: 1 items, 3) Satisfaction concerning the service: 3 items and 4) Overall satisfaction with support in management of sunitinib treatment: 1 item. Each item had 5 responses: very satisfied, satisfied, not very satisfied, not satisfied and no opinion. In this outcome measure number of participants who were either "Satisfied" or "Very Satisfied" for overall satisfaction were reported.
Time Frame: At the end of the study (At Month 6)
Population: Analysis population included all participants who were investigated by the doctors, who met the study eligibility criteria, had received at least 1 dose of Sunitinib and who were followed up by call center and completed a self-administered satisfaction questionnaire about management by call center.
Measure: Count of Participants; unit: Participants
Arm/Group | Call Center
Number analyzed (Participants) | 22
Participants | 19

19. Secondary Outcome: Mean Scores for Each Dimension on the Physician's Satisfaction (With the Management By the Telephone Call Center) Questionnaire
Description: Physician's satisfaction with call center service for participants' follow-up was assessed via the self-administered questionnaire completed at the end of the study. Questionnaire evaluated 3 dimensions with total of 5 items. Dimensions were: 1) Satisfaction concerning advice: had 3 items, 2) Satisfaction concerning management: 1 items and 3) Overall satisfaction: 1 item. Each item had 5 responses: very satisfied, satisfied, not very satisfied, not satisfied and no opinion equivalent to score of +2, +1, 1, -2 and no score respectively. A score was calculated for each dimension by calculating the mean scores obtained for each item if at least 50% of the items for the dimension have been completed (and are not "no opinion"). Overall possible mean score range for each dimension was +2 to -2, where higher scores signified higher satisfaction.
Time Frame: At the end of the study (At Month 6)
Population: Analysis population included all investigating doctors/physicians who completed a satisfaction questionnaire to assess the management of follow-up of participants by the call center. For this outcome measure 'Participant' refers to 'investigating physician'.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Physicians: Physicians who were investigating the participants being followed up by call center along with conventional method in the study.
Arm/Group | Physicians
Number analyzed (Participants) | 12
Units on a scale
  Satisfaction with the advice | 0.4 (1.1)
  Satisfaction with care | -0.6 (1.2)
  Overall satisfaction of participant care | 0.1 (1.4)

20. Secondary Outcome: Number of Investigating Physicians Who Reported Themselves Being "Satisfied" or "Very Satisfied" With the Management By the Telephone Call Center
Description: Physicians' satisfaction with call center service for participants' follow-up was assessed via the self-administered questionnaire completed at the end of the study. Questionnaire evaluated 3 dimensions with total of 5 item. Dimensions were: 1) Satisfaction concerning advice: had 3 items, 2) Satisfaction concerning management: 1 items and 3) Overall satisfaction: 1 item. Each item had 5 responses: very satisfied, satisfied, not very satisfied, not satisfied and no opinion. In this outcome measure number of physicians who were either "Satisfied" or "Very Satisfied" for overall satisfaction were reported.
Time Frame: Baseline up to 6 months
Population: as for outcome 19
Measure: Number; unit: Physicians
Arm/Group | Physicians
Number analyzed (Participants) | 12
Physicians | 7

21. Secondary Outcome: Total Number of Calls (Planned and Unplanned)
Description: 1 participant can call more than once during the study.
Time Frame: Baseline up to 6 months
Population: Analysis population included all participants who were investigated by the doctors, who met the study eligibility criteria, had received at least 1 dose of Sunitinib and who had telephone calls with call center. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number; unit: Calls
Arm/Group | Call Center
Number analyzed (Participants) | 35
Calls | 431

22. Secondary Outcome: Number of Participants Who Were Taking Sunitinib as Told to Call Center During the First Call
Description: Participants were followed up for taking their medication and they were supposed to respond either "yes" or "no". In this outcome measure participants who responded "Yes" are reported.
Time Frame: First call made anytime from baseline up to 6 months
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Call Center
Number analyzed (Participants) | 35
Participants | 33

23. Secondary Outcome: Number of Participants With Their Responses as "Yes" Against the Actions of Investigating Physicians, as Told to Call Center During the First Call
Description: Actions of investigating doctors/physicians: did doctor clearly explained how to take treatment, were participants given documentation about treatment by doctor or medical team, did doctor explained how to manage any side effects due to treatment which could occur and were prescriptions or orders for supportive medical treatments given by doctor. Participants responded either "Yes" or "No". In this outcome measure participants who responded "Yes" to each action are reported.
Time Frame: First call made anytime from baseline up to 6 months
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Call Center
Number analyzed (Participants) | 35
Participants
  Doctor clearly explained how to take treatment | 31
  Participants given documentation about treatment | 31
  Doctor explain manage side effect due to treatment | 27
  Prescriptions for supportive medical treatments | 27

24. Secondary Outcome: Number of Telephone Calls Describing Actions Taken by Call Center
Description: In this outcome measure number of telephone calls against each action taken/or described by the call center to the participants are reported. Actions taken by the call center included: 1) Given advice about managing the treatment: a) advice about taking Sunitinib, b) advice about using the Sunitinib follow-up diary, c) reporting any AE; 2) Given general preventative advice: a) advice about taking preventative systemic treatments, b) lifestyle advice, c) food/dietetic advice, d) oro-dental hygiene advice; 3) Given specific preventative advice for a type of AE: a) prevention of skin toxicities, b) prevention of gastrointestinal disorders, c) prevention of cardiac disorders, d) prevention of infectious/inflammatory problems, e)other preventative advice; 4) Actions recommended to participant: a) do not forget the planned consultation with the oncologist, b) get the additional investigations requested performed.
Time Frame: Baseline up to 6 months
Population: as for outcome 21
Measure: Number; unit: Telephone calls
Units Other Than Participants: Telephone calls
Arm/Group | Call Center
Number analyzed (Participants) | 35
Number analyzed (Telephone calls) | 431
Telephone calls
  Advice about managing treatment: taking Sunitinib | 266
  Advice about managing treatment:Sunitinib followup | 281
  Advice about managing treatment: Reporting any AE | 341
  General preventative advice: taking treatments | 263
  General preventative advice: Lifestyle advice | 278
  General preventative advice: Food/dietetic advice | 222
  General preventative advice: Orodental hygiene | 272
  Specific advice for type of AE: skin toxicities | 270
  Specific advice for type of AE: GI disorders | 271
  Specific advice for type of AE: cardiac disorders | 317
  Specific advice for type of AE: infectious problem | 233
  Specific advice for type of AE:preventative advice | 289
  Actions to participants:Do not forget consultation | 134
  Actions to participants: additional investigation | 137

25. Secondary Outcome: Number of Telephone Calls Where Participants Declared Adverse Events
Description: In this outcome measure total number of telephone calls where participants declared of any AE are reported. Participants could call more than once to declare AE.
Time Frame: Baseline up to 6 months
Population: Call center full analysis set (FAS) population included all participants who were investigated by doctors, who met the study eligibility criteria and had received at least 1 dose of Sunitinib and were followed up by call center. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number; unit: Telephone calls
Units Other Than Participants: Telephone calls
Arm/Group | Call Center
Number analyzed (Participants) | 35
Number analyzed (Telephone calls) | 431
Telephone calls | 280

ADVERSE EVENTS:
Time Frame: Baseline up to 6 months
Description: Same event may appear as AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study.
Arm/Group | Call Center | Standard of Care
All-Cause Mortality (participants affected / at risk) | 2/42 | 3/27
Serious Adverse Events (participants affected / at risk) | 12/42 | 15/27
Other Adverse Events (participants affected / at risk) | 42/42 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Call Center (N=42) | Standard of Care (N=27)
Anaemia (Blood and lymphatic system disorders) | 0 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Cardiac Failure (Cardiac disorders) | 1 | 0
Adrenal Insufficiency (Endocrine disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 1
Death (General disorders) | 1 | 0
General Physical Health Deterioration (General disorders) | 1 | 1
General Symptom (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Anti-Platelet Antibody Positive (Investigations) | 0 | 1
Weight Decreased (Investigations) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Aphasia (Nervous system disorders) | 0 | 1
Cerebral Haematoma (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 2 | 0
Clonus (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 0 | 1
Paralysis (Nervous system disorders) | 0 | 1
Sensorimotor Disorder (Nervous system disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 2
Renal Failure (Renal and urinary disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Call Center (N=42) | Standard of Care (N=27)
Anaemia (Blood and lymphatic system disorders) | 5 | 2
Blood Disorder (Blood and lymphatic system disorders) | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 12 | 1
Platelet Disorder (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 5
Tachycardia (Cardiac disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 5 | 0
Endocrine Disorder (Endocrine disorders) | 1 | 1
Hypothyroidism (Endocrine disorders) | 8 | 4
Conjunctivitis (Eye disorders) | 1 | 1
Dark Circles Under Eyes (Eye disorders) | 2 | 0
Eyelid Oedema (Eye disorders) | 4 | 0
Lacrimation Increased (Eye disorders) | 4 | 0
Abdominal Distension (Gastrointestinal disorders) | 5 | 0
Abdominal Pain (Gastrointestinal disorders) | 9 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 8 | 3
Anal Inflammation (Gastrointestinal disorders) | 2 | 1
Anorectal Disorder (Gastrointestinal disorders) | 2 | 0
Aphthous Ulcer (Gastrointestinal disorders) | 12 | 1
Cheilitis (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 7 | 1
Diarrhoea (Gastrointestinal disorders) | 24 | 5
Dry Mouth (Gastrointestinal disorders) | 10 | 2
Dyspepsia (Gastrointestinal disorders) | 11 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 0
Eructation (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 4 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 4 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 10 | 2
Gingival Pain (Gastrointestinal disorders) | 1 | 1
Gingivitis (Gastrointestinal disorders) | 13 | 0
Glossitis (Gastrointestinal disorders) | 5 | 0
Glossodynia (Gastrointestinal disorders) | 4 | 0
Haemorrhoids (Gastrointestinal disorders) | 4 | 1
Lip Pain (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 24 | 4
Oral Pain (Gastrointestinal disorders) | 2 | 0
Proctalgia (Gastrointestinal disorders) | 2 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 4 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 3
Toothache (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 15 | 3
Asthenia (General disorders) | 22 | 15
Chest Pain (General disorders) | 3 | 0
Chills (General disorders) | 6 | 0
Fatigue (General disorders) | 26 | 4
General Physical Health Deterioration (General disorders) | 2 | 0
General Symptom (General disorders) | 0 | 3
Inflammation (General disorders) | 2 | 0
Irritability (General disorders) | 3 | 0
Mucosal Dryness (General disorders) | 2 | 0
Mucosal Inflammation (General disorders) | 16 | 10
Oedema (General disorders) | 3 | 0
Oedema Peripheral (General disorders) | 5 | 0
Pain (General disorders) | 7 | 1
Pyrexia (General disorders) | 6 | 2
Xerosis (General disorders) | 3 | 0
Hepatocellular Injury (Hepatobiliary disorders) | 2 | 1
Jaundice (Hepatobiliary disorders) | 0 | 2
Hypersensitivity (Immune system disorders) | 1 | 1
Infection (Infections and infestations) | 4 | 2
Urinary Tract Infection (Infections and infestations) | 1 | 1
Blood Albumin Abnormal (Injury, poisoning and procedural complications) | 1 | 1
Blood Creatinine Increased (Injury, poisoning and procedural complications) | 5 | 1
Blood Lactate Dehydrogenase (Injury, poisoning and procedural complications) | 1 | 1
Blood Pressure Increased (Injury, poisoning and procedural complications) | 0 | 2
Blood Thyroid Stimulating Hormone Decreased (Injury, poisoning and procedural complications) | 0 | 2
Blood Thyroid Stimulating Hormone Increased (Injury, poisoning and procedural complications) | 6 | 5
Liver Function Test Abnormal (Injury, poisoning and procedural complications) | 1 | 1
Prothrombin Time Ratio (Injury, poisoning and procedural complications) | 2 | 0
Weight Decreased (Injury, poisoning and procedural complications) | 15 | 1
White Blood Cell Count Decreased (Injury, poisoning and procedural complications) | 1 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 27 | 7
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Bone Pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 6 | 0
Dysgeusia (Nervous system disorders) | 27 | 5
Headache (Nervous system disorders) | 15 | 3
Hyperaesthesia (Nervous system disorders) | 2 | 1
Neuropathy Peripheral (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 3 | 0
Depression (Psychiatric disorders) | 2 | 0
Food Aversion (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 4 | 0
Chromaturia (Renal and urinary disorders) | 3 | 0
Dysuria (Renal and urinary disorders) | 3 | 1
Proteinuria (Renal and urinary disorders) | 3 | 1
Renal Failure (Renal and urinary disorders) | 0 | 2
Balanitis (Reproductive system and breast disorders) | 2 | 0
Scrotal Erythema (Reproductive system and breast disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal Obstruction (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 10 | 2
Erythema (Skin and subcutaneous tissue disorders) | 8 | 0
Hair Colour Changes (Skin and subcutaneous tissue disorders) | 3 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 1
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 13 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 2
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 | 2
Skin Chapped (Skin and subcutaneous tissue disorders) | 2 | 0
Skin Discolouration (Skin and subcutaneous tissue disorders) | 9 | 0
Skin Fissures (Skin and subcutaneous tissue disorders) | 2 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 6 | 0
Skin Reaction (Skin and subcutaneous tissue disorders) | 3 | 1
Yellow Skin (Skin and subcutaneous tissue disorders) | 11 | 4
Tooth Extraction (Surgical and medical procedures) | 2 | 0
Hot Flush (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 33 | 10
Hypotension (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/42/NCT02187042/SAP_000.pdf
  • Study Protocol (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT02187042/Prot_001.pdf